CLINICAL TRIAL: NCT00962052
Title: Biomarker Discovery and Application in Bladder Cancer: Identification and Detection of Gene Methylation, Tumor Specific Antigenes Markers of BCG Treatment.
Brief Title: Biomarker Discovery and Application in Bladder Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wolfson Medical Center (Other Government)
Collaborators: Medical Diagnostic Laboratories, LLC (Industry)
Responsible Party: Prof Ami Sidi, Wolfson M.C
Other Study IDs: MDL0806
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, first void urine, bladder tumors and healthy tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators' long-term objective is to research and develop innovative new tests which diagnostic laboratories can use to 1) detect methylated DNA targets, 2) tumor specific antigens, and 3) markers of Bacillus Calmette-Guerin (BCG) treatment in patient urine samples. The investigators plan to detect methylated DNA targets and control targets by methylation-specific polymerase chain reaction (msPCR) on DNA isolated from urine samples from bladder cancer positive and negative patients to determine its sensitivity and specificity in detecting bladder cancer. The investigators plan to use patient sera as a tool to detect tumor specific antigens expressed by bladder cancer cell lines. Once a bladder tumor specific protein is identified, the investigators will assess its presence in the urine of bladder cancer patients and absence in healthy patients by enzyme-linked immunosorbent assay (ELISA). The investigators plan to use both in vitro models and patient clinical samples to elucidate the role of bladder epithelial cells in mediating BCG immunotherapy and identify biomarkers of treatment effectiveness. Once a biomarker is identified, the investigators will assess its presence in the urine of bladder cancer and absence in healthy patients.

Once the investigators determine the feasibility of these tests, the investigators will further perform an extensive clinical study, comparing the tests to existing diagnostic methods. This study will provide the foundation for FDA approval, which is required for tests to become widely accepted tools for clinicians to use in bladder cancer diagnosis. The investigators' tests will improve early detection of bladder cancer, thereby improving patient health and decrease cancer deaths, a key mission of the National Institutes of Health.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old

Exclusion Criteria:

* No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Those currently diagnosed and undergoing treatment for bladder cancer (100).
  2. Those currently diagnosed with other urogenital cancers including prostate cancer and kidney cancer (50).
  3. Those currently diagnosed with non-malignant urogenital conditions including urinary tract infection, interstitial cystitis, and kidney stones for specificity analysis (50).
  4. Healthy control patients (50).
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-12 (Estimated); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Wolfson Medical Center, Holon, Israel